CLINICAL TRIAL: NCT01383057
Title: Clear Corneal Incisions and Arcuate Incisions Utilizing FemtoSecond Laser Technology for Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEMTO 2011-2
Record Dates: First submitted 2011-06-24; First posted 2011-06-28 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Femtosecond Laser (Experimental)
  Interventions: Procedure: Femtosecond Laser

INTERVENTIONS:
Procedure: Femtosecond Laser — Using the Femtosecond Laser to make a clear corneal incision.

SUMMARY:
The purpose of this study is to prove the efficacy and safety of the Femtosecond laser to create a clear corneal incision during cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Study participants must have a cataract for which phacoemulsification extraction and posterior IOL implantation has been planned in at least one eye.
* Study participants should be capable of achieving better than 20/30 Snellen best corrected distance vision after cataract extraction and IOL implantation.

  * The surgeon may use the Mentor Potential Acuity Meter (PAM) laser interferometer, McIntyre Pinhole, or his/her judgment to estimate the patient's potential acuity.

Exclusion Criteria:

* Concurrent participation or participation in the last thirty days in any other clinical trial.
* Known steroid IOP responder
* Taking medications that may affect vision, IOP or ease of cataract surgery (e.g., Flomax, Glaucoma mediations, etc.)
* Acute or chronic disease or illness that would increase risk or confound study results (e.g., uncontrolled diabetes mellitus, immunocompromised, etc.)
* Uncontrolled systemic or ocular disease
* Corneal abnormalities (e.g., stromal, epithelial or endothelial dystrophies)
* Pseudoexfoliation
* Ocular hypertension IOP >25 mmHg by tonometry or glaucomatous changes in the optic nerve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure | 3 months
  Measure the fluid pressure inside the eye
Uncorrected and Best corrected Visual Acuity | one month
  Vision obtained with the best possible lens correction (Best corrected). Vision obtained without the use of glasses or contact lenses (Uncorrected).

CONTACTS AND LOCATIONS:
Locations (1):
- Loden Vision Centers, Goodlettsville, Tennessee, United States